CLINICAL TRIAL: NCT04026009
Title: A Phase I, Single-center, Randomized, Observer-blind, Placebo-controlled Study to Evaluate Safety, Reactogenicity and Immunogenicity of GSK's Clostridium Difficile Investigational Vaccine Based on the F2 Antigen With or Without AS01B Adjuvant, When Administered Intramuscularly According to a 0, 1-month Schedule to Healthy Adults Aged Between 18-45 Years and Between 50-70 Years, Followed by an Additional Dose Administered in a Partial Blind Manner Within an Interval of Approximately 15 Months After Dose 2, in a Subcohort of Subjects Aged 50-70 Years
Brief Title: Safety and Immunogenicity Study of GSK's Clostridium Difficile Vaccine 2904545A When Administered in Healthy Adults Aged 18-45 Years and 50-70 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 208109; 2018-002304-14 (EudraCT Number)
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Clostridium Infections
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: A 4-step staggered design will be used to ensure maximum safety of the participating subjects:
  Step 1: Vaccination of approximately 20 subjects aged 18-45 years. Step 2: Vaccination of approximately 20 subjects aged 50-70 years. Step 3: Vaccination of approximately 30 subjects aged 50-70 years. An iSRC will review all accumulating safety data after Dose 1 and 2 in Steps 1 to 3. If considered appropriate to proceed, the next step will start.
  Step 4: Vaccination of approximately 70 subjects aged 50-70 years. An iSRC will review all accumulating safety data 3 weeks after the start of vaccination in Step 4 and then about every 3 weeks until all subjects have received Dose 1. In addition, the iSRC will review all safety data after Dose 2 and after that a subcohort of subjects will receive the third dose. If there are any safety concerns observed during SRT reviews post Dose 3, an ad hoc iSRC meeting will take place to review the unblinded safety data.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, observer-blind and partial blind (only for third dose) study.
  Given the different appearance of the C.difficile investigational vaccines and placebo, double blinding is not possible, and the study will be conducted in an observer-blind manner. In an observer-blind study, the subject, the Contract Research Organization personnel, and the study center and Sponsor personnel involved in the clinical evaluation of the subjects are blinded while other study personnel may be aware of the treatment assignment.
  When all data up to Day 61 are available, a statistical analysis will be performed.This analysis may lead to the unblinding of some subjects.A statistician will be unblinded for the analysis.The study will be considered as partial blind from this point onwards.
  The Investigator and the subjects will not have access to the treatment allocation up to Day 390. After Day 390, only the subjects will remain fully blinded, while the Investigator will be partially blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CDIFF Ag 18 - 45 Years Group (Experimental): Healthy male and female subjects, aged between and including 18 and 45 years old, who receive CDIFF antigen (Ag) vaccine administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule.
  Interventions: Biological: C. difficile investigational vaccine based on the F2 antigen (GSK2904545A)
- Placebo 18 - 45 Years Group (Placebo Comparator): Healthy male and female subjects, aged between and including 18 and 45 years old, who receive Placebo administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule.
  Interventions: Drug: Placebo
- CDIFF Ag 50 - 70 Years Group (Experimental): Healthy male and female subjects, aged between and including 50 and 70 years old, who receive CDIFF antigen (Ag) vaccine administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule. A third dose of CDIFF Ag vaccine is to be administered to a subcohort of subjects aged 50-70 years, approximately 15 months after the administration of the second dose.
  Interventions: Biological: C. difficile investigational vaccine based on the F2 antigen (GSK2904545A)
- CDIFF Ag + AS01B 50 - 70 Years Group (Experimental): Healthy male and female subjects, aged between and including 50 and 70 years old, who receive CDIFF Ag + AS01B adjuvant vaccine administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule. A third dose of CDIFF Ag + AS01B adjuvant vaccine is to be administered to a subcohort of subjects aged 50-70 years, approximately 15 months after the administration of the second dose.
  Interventions: Biological: C. difficile investigational vaccine based on the F2 antigen (GSK2904545A) adjuvanted with AS01B
- Placebo 50 - 70 Years Group (Placebo Comparator): Healthy male and female subjects, aged between and including 50 and 70 years old, who receive Placebo administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: C. difficile investigational vaccine based on the F2 antigen (GSK2904545A) — Subjects in CDIFF Ag 18 - 45 Years and CDIFF Ag 50 - 70 Years Groups will receive 2 or 3 doses (0.5 mL each) of CDIFF Ag vaccine.
  The vaccine will be administered intramuscularly in the deltoid, at a 0, 1-month dose interval. The third dose will be administered approximately 15 months after the second dose.
  Other Names: CDIFF Ag
  Arms: CDIFF Ag 18 - 45 Years Group; CDIFF Ag 50 - 70 Years Group
Biological: C. difficile investigational vaccine based on the F2 antigen (GSK2904545A) adjuvanted with AS01B — Subjects in CDIFF Ag + AS01B 50 - 70 Years Group will receive 2 or 3 doses (0.5 mL each) of CDIFF Ag + AS01B vaccine.
  The vaccine will be administered intramuscularly in the deltoid, at a 0, 1-month dose interval. The third dose will be administered approximately 15 months after the second dose.
  Other Names: CDIFF Ag + AS01B
  Arms: CDIFF Ag + AS01B 50 - 70 Years Group
Drug: Placebo — Subjects will receive 2 doses (0.5 mL each) of Placebo, administered intramuscularly in the deltoid, at a 0, 1-month dose interval.
  Arms: Placebo 18 - 45 Years Group; Placebo 50 - 70 Years Group

SUMMARY:
The purpose of this study is to generate safety, reactogenicity (assessment of any expected or unexpected side effect of the vaccine) and immunogenicity (ability to induce an immune response) data for the development of a candidate Clostridium difficile (C. difficile) vaccine that would protect against primary cases of Clostridium difficile infection (CDI) and CDI recurrence.

Clostridium difficile infection is a major cause of gastrointestinal illness with approximately 500,000 infections and the leading cause of gastroenteritis associated death with 29,000 deaths annually in the United States of America (USA). The emergence of extremely infectious varieties/types of C. difficile has contributed to increase the number and severity of CDI cases. In recent years, some countries (United Kingdom) have implemented hospital hygiene and other measures which resulted in significant reductions in the number of cases. The burden is, however, expected to remain significant until vaccination is available.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who, in the opinion of the Investigator, can and will comply with the requirements of the protocol.
2. Written or witnessed/thumb print informed consent obtained from the subject prior to performance of any study specific procedure.
3. For Step 1 only: A male or female between, and including, 18-45 years of age at the time of the first vaccination.
4. For Steps 2, 3, and 4: A male or female between, and including, 50-70 years of age at the time of the first vaccination.
5. Healthy subjects as established by medical history and clinical examination before entering into the study.
6. Subjects free of any uncontrolled chronic illnesses as established by medical history and clinical examination before entering into the study.
7. Female subjects of non-childbearing potential may be enrolled in the study.

   * Non-childbearing potential is defined as premenarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy, or post-menopause.

Female subjects of childbearing potential may be enrolled in the study, if the subject:

* Has practiced adequate contraception for 30 days prior to vaccination, and
* Has a negative urine pregnancy test on the day of vaccination, and
* Has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

1. Health condition that, in the opinion of the Investigator, may interfere with optimal participation in the study or place the volunteer at increased risk of AEs. Study clinicians, in consultation with the Principal Investigator will use clinical judgment on a case by case basis to assess safety risks under this criterion. The Principal Investigator will consult with the Medical Monitor as appropriate.
2. Use of any investigational or nonregistered product other than the study vaccine(s) during the period starting 30 days before the first dose of study vaccine(s) (Day 29 to Day 1), or planned use during the study period.
3. Any medical condition that in the judgment of the Investigator would make IM injection unsafe and subjects under treatment with anticoagulant therapy.
4. Chronic administration of immunosuppressants or other immune modifying drugs during the period starting 3 months prior to the first vaccination. For corticosteroids, this will mean prednisone ≥ 5 milligrams per day (mg/day) (for adult subjects), or equivalent. Inhaled and topical steroids are allowed.
5. Administration of long acting immune modifying drugs at any time during the study period.
6. Administration of immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation or autoimmune disease.
7. Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first vaccination of study treatment or planned administration during the study period.
8. Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 6 weeks before the first vaccination and ending 6 weeks after the last vaccination, with the exception of inactivated influenza vaccine which can be administered up to 14 days before or from 30 days after the last study vaccination.

   In case an emergency mass vaccination for an unforeseen public health threat (eg, a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if, necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.
9. Planned administration of GSK's Herpes Zoster vaccine marketed as Shingrix or an adjuvanted recombinant varicella zoster virus envelope gE subunit vaccine (HZ/su) within 180 days before the first dose and within 180 days after the last dose of the study vaccine.
10. Planned elective surgery during the study period.
11. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
12. Body mass index < 19 kg/m^2 or ≥ 35 kg/m^2.
13. Clinically relevant physical examination abnormalities.
14. For subjects aged 18 - 45 years, Grade 2 or higher abnormal hematological, biochemical, and urinary parameters.
15. For subjects aged 50 - 70 years, Grade 3 or higher abnormal hematological, biochemical, and urinary parameters.
16. Documentation of current or prior episode of CDI.
17. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
18. Recurrent history or uncontrolled neurological disorders or seizures.
19. Family history of congenital or hereditary immunodeficiency.
20. History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
21. Acute disease and/or fever at the time of enrollment.

    * Fever is defined as temperature ≥ 38.0°C/100.4°F. The preferred location for measuring temperature in this study will be the oral cavity.
    * Subjects with a minor illness, without fever, may be enrolled at the discretion of the Investigator.
22. Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
23. Pregnant or lactating female.
24. History of intestinal bleeding or history of diverticular intestinal bleeding.
25. Surgery for gastrointestinal malignancy in the period starting 3 months prior to the first vaccination.
26. History of chronic alcohol consumption and/or drug abuse as deemed by the Investigator to render the potential subject unable/unlikely to provide accurate safety reports.
27. Female planning to become pregnant or planning to discontinue contraceptive precautions.
28. Documented human immunodeficiency virus positive subject, known positivity for the surface antigen of the hepatitis B virus or known positive serologic test for the hepatitis C virus.
29. Involvement in the planning and/or conduct of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Leroux-Roels I, Alhatemi A, Caubet M, De Boever F, de Wergifosse B, El Idrissi M, Ferreira GS, Jacobs B, Lambert A, Morel S, Servais C, Yarzabal JP. Safety and Immunogenicity of an Adjuvanted Clostridioides difficile Vaccine Candidate in Healthy Adults: A Randomized Placebo-Controlled Phase 1 Study. J Infect Dis. 2025 Mar 17;231(3):e511-e520. doi: 10.1093/infdis/jiae466. PMID 39447053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in this study were randomized in 5 groups on 2 age categories. After study interventions, as pre-assigned in protocol, the participants were followed up for safety, reactogenicity, and immunogenicity analysis until the end of the study.
Groups:
- CDIFF Ag 50 - 70 Years Group: Healthy male and female subjects, aged between and including 50 and 70 years old, who receive CDIFF antigen (Ag) vaccine administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule. A third dose of CDIFF Ag vaccine was administered to a set of participants in this group, approximately 15 months after the administration of the second dose.
- CDIFF Ag + AS01B 50 - 70 Years Group: Healthy male and female subjects, aged between and including 50 and 70 years old, who receive CDIFF Ag + AS01B adjuvant vaccine administered intramuscularly in the deltoid, according to a 0, 1-month vaccination schedule. A third dose of CDIFF Ag + AS01B adjuvant vaccine was administered to a set of participants in this group, approximately 15 months after the administration of the second dose.
Period: Overall Study
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Started | 10 | 10 | 45 | 45 | 30
Completed | 10 | 10 | 45 | 44 | 29
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 0 | 1 | 0
Not completed — Consent withdrawal, not due to adverse event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group | Total
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (6.8) | 31.5 (7.7) | 60.7 (6.1) | 60.8 (6.0) | 58.9 (6.2) | 56.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 30 | 30 | 20 | 90
  Male | 5 | 5 | 15 | 15 | 10 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 10 | 45 | 45 | 30 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, After Each Vaccine Dose
Description: Assessed solicited local symptoms are pain at injection site, redness at injection site and swelling at injection site.
  Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, pain that pre-vents normal every day activities. Grade 3 redness/swelling = redness/swelling with a maximum diameter greater (>) than 100 millimeters (mm).
Time Frame: During the 7-day follow-up period (from the day of vaccination up to 6 subsequent days) after each vaccination
Population: The analysis is performed on the Solicited Safety Set, which included all subjects who received at least one dose of the study vaccine and for whom solicited safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants
  Any Erythema, after Dose 1 | 0 | 0 | 0 | 8 | 0
  Grade 3 Erythema, after Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Pain, after Dose 1 | 0 | 1 | 0 | 40 | 1
  Grade 3 Pain, after Dose 1 | 0 | 0 | 0 | 1 | 0
  Any Swelling, after Dose 1 | 0 | 0 | 0 | 3 | 0
  Grade 3 Swelling, after Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Erythema, after Dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Erythema, after Dose 2 | 0 | 0 | 0 | 19 | 0
  Grade 3 Erythema, after Dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Erythema, after Dose 2 | 0 | 0 | 0 | 4 | 0
  Any Pain, after Dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Pain, after Dose 2 | 2 | 1 | 2 | 38 | 0
  Grade 3 Pain, after Dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Pain, after Dose 2 | 0 | 0 | 0 | 1 | 0
  Any Swelling, after Dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Swelling, after Dose 2 | 0 | 0 | 0 | 4 | 0
  Grade 3 Swelling, after Dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 2
  Grade 3 Swelling, after Dose 2 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3, Related and Grade 3 Related Solicited General Symptoms, After Each Vaccine Dose
Description: Assessed solicited general symptoms are fatigue, fever [defined as oral temperature equal to or higher than (>=) 38 degrees Celsius (°C)], gastrointestinal symptoms (nausea, vomiting, diarrhea, and/or abdominal pain), headache, myalgia, shivering and arthralgia.
  Any = occurrence of the symptom regardless of intensity grade and relationship to vaccination. Grade 3 symptom = symptom that prevents normal, everyday activities. Grade 3 fever = oral temperature higher (>) than 39.0°C. Related symptom = symptom assessed by the investigator as causally related to the study vaccination. Grade 3 related symptom = Grade 3 symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day follow-up period (from the day of vaccination up to 6 subsequent days) after each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants
  Any Arthralgia, after dose 1 | 0 | 0 | 0 | 5 | 3
  Grade 3 Arthralgia, after dose 1 | 0 | 0 | 0 | 0 | 0
  Related Arthralgia, after dose 1 | 0 | 0 | 0 | 4 | 3
  Grade 3 related Arthralgia, after dose 1 | 0 | 0 | 0 | 0 | 0
  Any Fatigue, after dose 1 | 4 | 2 | 9 | 20 | 7
  Grade 3 Fatigue, after dose 1 | 0 | 0 | 0 | 0 | 1
  Related Fatigue, after dose 1 | 2 | 1 | 8 | 19 | 7
  Grade 3 related Fatigue, after dose 1 | 0 | 0 | 0 | 0 | 1
  Any Gastrointestinal symptoms, after dose 1 | 1 | 3 | 8 | 7 | 5
  Grade 3 Gastrointestinal symptoms, after dose 1 | 1 | 1 | 0 | 0 | 0
  Related Gastrointestinal symptoms, after dose 1 | 1 | 2 | 5 | 7 | 3
  Grade 3 related Gastrointestinal symptoms, after dose 1 | 1 | 1 | 0 | 0 | 0
  Any Headache, after dose 1 | 2 | 2 | 12 | 18 | 6
  Grade 3 Headache, after dose 1 | 0 | 0 | 0 | 0 | 0
  Related Headache, after dose 1 | 1 | 1 | 9 | 16 | 6
  Grade 3 related Headache, after dose 1 | 0 | 0 | 0 | 0 | 0
  Any Myalgia, after dose 1 | 1 | 1 | 3 | 7 | 3
  Grade 3 Myalgia, after dose 1 | 0 | 0 | 0 | 0 | 0
  Related Myalgia, after dose 1 | 1 | 0 | 2 | 7 | 3
  Grade 3 related Myalgia, after dose 1 | 0 | 0 | 0 | 0 | 0
  Any Shivering, after dose 1 | 0 | 0 | 3 | 5 | 4
  Grade 3 Shivering, after dose 1 | 0 | 0 | 0 | 0 | 1
  Related Shivering, after dose 1 | 0 | 0 | 3 | 5 | 4
  Grade 3 related Shivering, after dose 1 | 0 | 0 | 0 | 0 | 1
  Any Temperature (C), after dose 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Temperature (C), after dose 1 | 0 | 0 | 0 | 0 | 0
  Related Temperature (C), after dose 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 related Temperature (C), after dose 1 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Arthralgia, after dose 2 | 0 | 1 | 4 | 9 | 2
  Grade 3 Arthralgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Arthralgia, after dose 2 | 0 | 0 | 0 | 0 | 0
  Related Arthralgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Arthralgia, after dose 2 | 0 | 1 | 3 | 9 | 0
  Grade 3 related Arthralgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Arthralgia, after dose 2 | 0 | 0 | 0 | 0 | 0
  Any Fatigue, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Fatigue, after dose 2 | 1 | 0 | 8 | 26 | 7
  Grade 3 Fatigue, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Fatigue, after dose 2 | 0 | 0 | 0 | 2 | 0
  Related Fatigue, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Fatigue, after dose 2 | 1 | 0 | 5 | 26 | 5
  Grade 3 related Fatigue, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Fatigue, after dose 2 | 0 | 0 | 0 | 2 | 0
  Any Gastrointestinal symptoms, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Gastrointestinal symptoms, after dose 2 | 0 | 0 | 3 | 12 | 1
  Grade 3 Gastrointestinal symptoms, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Gastrointestinal symptoms, after dose 2 | 0 | 0 | 0 | 0 | 0
  Related Gastrointestinal symptoms, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Gastrointestinal symptoms, after dose 2 | 0 | 0 | 3 | 11 | 1
  Grade 3 related Gastrointestinal symptoms, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Gastrointestinal symptoms, after dose 2 | 0 | 0 | 0 | 0 | 0
  Any Headache, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Headache, after dose 2 | 1 | 1 | 8 | 19 | 6
  Grade 3 Headache, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Headache, after dose 2 | 1 | 0 | 0 | 1 | 0
  Related Headache, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Headache, after dose 2 | 0 | 1 | 6 | 19 | 6
  Grade 3 related Headache, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Headache, after dose 2 | 0 | 0 | 0 | 1 | 0
  Any Myalgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Myalgia, after dose 2 | 2 | 0 | 4 | 19 | 1
  Grade 3 Myalgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Myalgia, after dose 2 | 0 | 0 | 0 | 0 | 0
  Related Myalgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Myalgia, after dose 2 | 2 | 0 | 2 | 18 | 0
  Grade 3 related Myalgia, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Myalgia, after dose 2 | 0 | 0 | 0 | 0 | 0
  Any Shivering, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Shivering, after dose 2 | 0 | 0 | 3 | 19 | 2
  Grade 3 Shivering, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Shivering, after dose 2 | 0 | 0 | 0 | 4 | 0
  Related Shivering, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Shivering, after dose 2 | 0 | 0 | 2 | 19 | 1
  Grade 3 related Shivering, after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Shivering, after dose 2 | 0 | 0 | 0 | 4 | 0
  Any Temperature (C), after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Any Temperature (C), after dose 2 | 0 | 0 | 0 | 5 | 0
  Grade 3 Temperature (C), after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 Temperature (C), after dose 2 | 0 | 0 | 0 | 0 | 0
  Related Temperature (C), after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Related Temperature (C), after dose 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 related Temperature (C), after dose 2: number analyzed (Participants) | 10 | 10 | 45 | 42 | 29
  Grade 3 related Temperature (C), after dose 2 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Any, Grade 3, Related, Grade 3 Related and Medically Attended Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is any adverse event reported in addition to those solicited during the clinical study. Also, any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
  Potential unsolicited AEs may be medically attended (defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider) or were of concern to the subjects.
  Any = occurrence of the symptom regardless of intensity grade and relationship to vaccination. Grade 3 symptom = symptom that prevents normal, everyday activities. Related symptom = symptom assessed by the investigator as causally related to the study vaccination. Grade 3 related symptom = Grade 3 symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 30-day follow-up period (from the day of vaccination up to 29 subsequent days) after any vaccination
Population: The analysis is performed on the Exposed Set, which included all subjects who received at least one dose of the study vaccine and for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants
  Any unsolicited AEs | 3 | 2 | 22 | 27 | 11
  Grade 3 unsolicited AEs | 1 | 0 | 2 | 3 | 1
  Related unsolicited AEs | 0 | 0 | 0 | 8 | 0
  Grade 3 related unsolicited AEs | 0 | 0 | 0 | 0 | 0
  Medically attended unsolicited AEs | 1 | 0 | 8 | 14 | 3

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, represents a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 up to and including Day 390 (Epoch 001)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants | 0 | 1 | 3 | 3 | 0

5. Primary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of adverse events of specific interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: During the whole study period (from Day 1 up to Day 390 [for subjects receiving 2 vaccine doses] and from Day 1 up to Day 670 [for subjects receiving 3 vaccine doses])
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants | 0 | 0 | 2 | 0 | 0

6. Primary Outcome: Number of Subjects With Hematological, Biochemical, and Urinary Laboratory Abnormalities at Screening
Description: Hematological (white blood cells, platelet count, hemoglobin level), biochemical (alanine aminotransferase, aspartate aminotransferase, creatinine, C-reactive protein and urate/uric acid) and urinary (protein, glucose and red blood cells) parameters are assessed. C-reactive protein is only assessed during the screening visit. Grades are based on the local laboratory normal ranges and derived from the FDA Toxicity Grading Scale for laboratory abnormalities.
Time Frame: At Screening (from Day -15 up to Day -1 [for subjects receiving 2 vaccine doses] and at Day 476 [for subjects receiving 3 vaccine doses])
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants
  Hemoglobin, at Screening (Below Normal Range) | 0 | 0 | 3 | 1 | 0
  Hemoglobin, at Screening (Above Normal Range) | 0 | 0 | 3 | 2 | 1
  Hemoglobin, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Hemoglobin, at Day 476 (Below Normal Range) |  |  | 1 | 0 | 0
  Hemoglobin, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Hemoglobin, at Day 476 (Above Normal Range) |  |  | 2 | 0 | 0
  White Blood Cells, at Screening (Below Normal Range) | 0 | 0 | 0 | 2 | 0
  White Blood Cells, at Screening (Above Normal Range) | 0 | 0 | 3 | 0 | 3
  White Blood Cells, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  White Blood Cells, at Day 476 (Below Normal Range) |  |  | 1 | 1 | 0
  White Blood Cells, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  White Blood Cells, at Day 476 (Above Normal Range) |  |  | 1 | 0 | 0
  Platelets, at Screening (Below Normal Range) | 1 | 1 | 0 | 2 | 0
  Platelets, at Screening (Above Normal Range) | 0 | 0 | 1 | 1 | 4
  Platelets, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Platelets, at Day 476 (Below Normal Range) |  |  | 1 | 1 | 0
  Platelets, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Platelets, at Day 476 (Above Normal Range) |  |  | 3 | 2 | 0
  Alanine Aminotransferase, at Screening (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Screening (Above Normal Range) | 0 | 0 | 2 | 8 | 4
  Alanine Aminotransferase, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Alanine Aminotransferase, at Day 476 (Below Normal Range) |  |  | 0 | 0 | 0
  Alanine Aminotransferase, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Alanine Aminotransferase, at Day 476 (Above Normal Range) |  |  | 1 | 2 | 0
  Aspartate Aminotransferase, at Screening (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Screening (Above Normal Range) | 0 | 0 | 0 | 4 | 1
  Aspartate Aminotransferase, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Aspartate Aminotransferase, at Day 476 (Below Normal Range) |  |  | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Aspartate Aminotransferase, at Day 476 (Above Normal Range) |  |  | 1 | 1 | 0
  Creatinine, at Screening (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Creatinine, at Screening (Above Normal Range) | 0 | 0 | 3 | 2 | 0
  Creatinine, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Creatinine, at Day 476 (Below Normal Range) |  |  | 0 | 0 | 0
  Creatinine, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Creatinine, at Day 476 (Above Normal Range) |  |  | 1 | 0 | 0
  Urate, at Screening (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Screening (Above Normal Range) | 1 | 0 | 6 | 9 | 5
  Urate, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Urate, at Day 476 (Below Normal Range) |  |  | 0 | 0 | 0
  Urate, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  Urate, at Day 476 (Above Normal Range) |  |  | 4 | 3 | 0
  C Reactive Protein, at Screening (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  C Reactive Protein, at Screening (Above Normal Range) | 2 | 1 | 1 | 3 | 4
  C Reactive Protein, at Day 476 (Below Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  C Reactive Protein, at Day 476 (Below Normal Range) |  |  | 0 | 0 | 0
  C Reactive Protein, at Day 476 (Above Normal Range): number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
  C Reactive Protein, at Day 476 (Above Normal Range) |  |  | 0 | 1 | 0

7. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 8
Description: Hematological (white blood cells, platelet count, hemoglobin level), biochemical (alanine aminotransferase, aspartate aminotransferase, creatinine and urate/uric acid) parameters are assessed. Grades are based on the local laboratory normal ranges and derived from the FDA Toxicity Grading Scale for laboratory abnormalities.
Time Frame: At Day 8
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 45 | 30
Participants
  Hemoglobin, at Day 8 (Below Normal Range) | 0 | 0 | 2 | 1 | 0
  Hemoglobin, at Day 8 (Above Normal Range) | 0 | 1 | 2 | 1 | 1
  White Blood Cells, at Day 8 (Below Normal Range) | 0 | 0 | 1 | 2 | 1
  White Blood Cells, at Day 8 (Above Normal Range) | 0 | 0 | 1 | 0 | 1
  Platelets, at Day 8 (Below Normal Range) | 1 | 1 | 1 | 2 | 1
  Platelets, at Day 8 (Above Normal Range) | 1 | 0 | 1 | 1 | 1
  Alanine Aminotransferase, at Day 8 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 8 (Above Normal Range) | 1 | 0 | 0 | 10 | 6
  Aspartate Aminotransferase, at Day 8 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 8 (Above Normal Range) | 0 | 0 | 0 | 3 | 2
  Creatinine, at Day 8 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Creatinine, at Day 8 (Above Normal Range) | 0 | 0 | 3 | 2 | 0
  Urate, at Day 8 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 8 (Above Normal Range) | 1 | 0 | 5 | 9 | 6

8. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 31
Description: as for outcome 7
Time Frame: At Day 31
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 43 | 29
Participants
  Hemoglobin, at Day 31 (Below Normal Range) | 0 | 0 | 2 | 3 | 0
  Hemoglobin, at Day 31 (Above Normal Range) | 0 | 1 | 2 | 0 | 1
  White Blood Cells, at Day 31 (Below Normal Range) | 0 | 0 | 0 | 0 | 1
  White Blood Cells, at Day 31 (Above Normal Range) | 1 | 0 | 0 | 0 | 0
  Platelets, at Day 31 (Below Normal Range) | 0 | 1 | 1 | 1 | 0
  Platelets, at Day 31 (Above Normal Range) | 0 | 0 | 1 | 1 | 0
  Alanine Aminotransferase, at Day 31 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 31 (Above Normal Range) | 0 | 1 | 2 | 8 | 4
  Aspartate Aminotransferase, at Day 31 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 31 (Above Normal Range) | 0 | 0 | 0 | 4 | 1
  Creatinine, at Day 31 (Below Normal Range) | 0 | 0 | 1 | 0 | 0
  Creatinine, at Day 31 (Above Normal Range) | 0 | 0 | 3 | 3 | 0
  Urate, at Day 31 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 31 (Above Normal Range) | 1 | 0 | 6 | 9 | 5

9. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 38
Description: as for outcome 7
Time Frame: At Day 38
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 43 | 28
Participants
  Hemoglobin, at Day 38 (Below Normal Range) | 0 | 0 | 0 | 2 | 1
  Hemoglobin, at Day 38 (Above Normal Range) | 0 | 0 | 3 | 1 | 1
  White Blood Cells, at Day 38 (Below Normal Range) | 0 | 0 | 0 | 0 | 2
  White Blood Cells, at Day 38 (Above Normal Range) | 0 | 0 | 1 | 1 | 1
  Platelets, at Day 38 (Below Normal Range) | 0 | 1 | 0 | 1 | 0
  Platelets, at Day 38 (Above Normal Range) | 0 | 0 | 2 | 1 | 1
  Alanine Aminotransferase, at Day 38 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 38 (Above Normal Range) | 1 | 1 | 1 | 8 | 3
  Aspartate Aminotransferase, at Day 38 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 38 (Above Normal Range) | 0 | 0 | 0 | 2 | 2
  Creatinine, at Day 38 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Creatinine, at Day 38 (Above Normal Range) | 0 | 0 | 2 | 1 | 1
  Urate, at Day 38 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 38 (Above Normal Range) | 1 | 0 | 9 | 9 | 5

10. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 180
Description: as for outcome 7
Time Frame: At Day 180
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 44 | 29
Participants
  Hemoglobin, at Day 180 (Below Normal Range) | 0 | 1 | 2 | 2 | 0
  Hemoglobin, at Day 180 (Above Normal Range) | 0 | 1 | 2 | 1 | 1
  White Blood Cells, at Day 180 (Below Normal Range) | 0 | 1 | 0 | 5 | 1
  White Blood Cells, at Day 180 (Above Normal Range) | 0 | 0 | 0 | 0 | 0
  Platelets, at Day 180 (Below Normal Range) | 1 | 1 | 1 | 2 | 0
  Platelets, at Day 180 (Above Normal Range) | 2 | 0 | 4 | 2 | 1
  Alanine Aminotransferase, at Day 180 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 180 (Above Normal Range) | 2 | 0 | 1 | 7 | 2
  Aspartate Aminotransferase, at Day 180 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 180 (Above Normal Range) | 1 | 0 | 0 | 2 | 2
  Creatinine, at Day 180 (Below Normal Range) | 0 | 0 | 1 | 0 | 0
  Creatinine, at Day 180 (Above Normal Range) | 0 | 0 | 2 | 1 | 0
  Urate, at Day 180 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 180 (Above Normal Range) | 0 | 0 | 5 | 9 | 5

11. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 390
Description: as for outcome 7
Time Frame: At Day 390
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 10 | 10 | 45 | 44 | 29
Participants
  Hemoglobin, at Day 390 (Below Normal Range) | 0 | 0 | 2 | 0 | 1
  Hemoglobin, at Day 390 (Above Normal Range) | 0 | 0 | 2 | 0 | 1
  White Blood Cells, at Day 390 (Below Normal Range) | 1 | 0 | 2 | 4 | 3
  White Blood Cells, at Day 390 (Above Normal Range) | 0 | 0 | 1 | 0 | 0
  Platelets, at Day 390 (Below Normal Range) | 1 | 1 | 1 | 2 | 0
  Platelets, at Day 390 (Above Normal Range) | 1 | 0 | 3 | 2 | 2
  Alanine Aminotransferase, at Day 390 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 390 (Above Normal Range) | 1 | 0 | 2 | 8 | 4
  Aspartate Aminotransferase, at Day 390 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 390 (Above Normal Range) | 0 | 1 | 1 | 2 | 2
  Urate, at Day 390 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 390 (Above Normal Range) | 1 | 0 | 6 | 7 | 5

12. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 476
Description: as for outcome 7
Time Frame: At Day 476
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 0 | 0 | 20 | 22 | 0
Participants
  Hemoglobin, at Day 476 (Below Normal Range) | 0 | 0 | 1 | 0 | 0
  Hemoglobin, at Day 476 (Above Normal Range) | 0 | 0 | 2 | 0 | 0
  White Blood Cells, at Day 476 (Below Normal Range) | 0 | 0 | 1 | 1 | 0
  White Blood Cells, at Day 476 (Above Normal Range) | 0 | 0 | 1 | 0 | 0
  Platelets, at Day 476 (Below Normal Range) | 0 | 0 | 1 | 1 | 0
  Platelets, at Day 476 (Above Normal Range) | 0 | 0 | 3 | 2 | 0
  Alanine Aminotransferase, at Day 476 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 476 (Above Normal Range) | 0 | 0 | 1 | 2 | 0
  Aspartate Aminotransferase, at Day 476 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 476 (Above Normal Range) | 0 | 0 | 1 | 1 | 0
  Creatinine, at Day 476 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Creatinine, at Day 476 (Above Normal Range) | 0 | 0 | 1 | 0 | 0
  Urate, at Day 476 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 476 (Above Normal Range) | 0 | 0 | 4 | 3 | 0

13. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 491
Description: as for outcome 7
Time Frame: At Day 491
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 0 | 0 | 20 | 20 | 0
Participants
  Hemoglobin, at Day 491 (Below Normal Range) | 0 | 0 | 1 | 1 | 0
  Hemoglobin, at Day 491 (Above Normal Range) | 0 | 0 | 2 | 0 | 0
  White Blood Cells, at Day 491 (Below Normal Range) | 0 | 0 | 3 | 2 | 0
  White Blood Cells, at Day 491 (Above Normal Range) | 0 | 0 | 1 | 0 | 0
  Platelets, at Day 491 (Below Normal Range) | 0 | 0 | 1 | 1 | 0
  Platelets, at Day 491 (Above Normal Range) | 0 | 0 | 2 | 2 | 0
  Alanine Aminotransferase, at Day 491 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 491 (Above Normal Range) | 0 | 0 | 1 | 3 | 0
  Aspartate Aminotransferase, at Day 491 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 491 (Above Normal Range) | 0 | 0 | 0 | 2 | 0
  Creatinine, at Day 491 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Creatinine, at Day 491 (Above Normal Range) | 0 | 0 | 1 | 0 | 0
  Urate, at Day 491 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 491 (Above Normal Range) | 0 | 0 | 4 | 4 | 0

14. Primary Outcome: Number of Subjects With Hematological and Biochemical Laboratory Abnormalities at Day 670
Description: as for outcome 7
Time Frame: At Day 670
Population: The analysis is performed on the Enrolled Set, which included all subjects who signed the Informed Consent Form (ICF).
Measure: Count of Participants; unit: Participants
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 0 | 0 | 20 | 20 | 0
Participants
  Hemoglobin, at Day 670 (Below Normal Range) | 0 | 0 | 2 | 1 | 0
  Hemoglobin, at Day 670 (Above Normal Range) | 0 | 0 | 2 | 0 | 0
  White Blood Cells, at Day 670 (Below Normal Range) | 0 | 0 | 2 | 2 | 0
  White Blood Cells, at Day 670 (Above Normal Range) | 0 | 0 | 1 | 1 | 0
  Platelets, at Day 670 (Below Normal Range) | 0 | 0 | 1 | 0 | 0
  Platelets, at Day 670 (Above Normal Range) | 0 | 0 | 2 | 2 | 0
  Alanine Aminotransferase, at Day 670 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase, at Day 670 (Above Normal Range) | 0 | 0 | 2 | 2 | 0
  Aspartate Aminotransferase, at Day 670 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, at Day 670 (Above Normal Range) | 0 | 0 | 1 | 1 | 0
  Creatinine, at Day 670 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Creatinine, at Day 670 (Above Normal Range) | 0 | 0 | 2 | 1 | 0
  Urate, at Day 670 (Below Normal Range) | 0 | 0 | 0 | 0 | 0
  Urate, at Day 670 (Above Normal Range) | 0 | 0 | 2 | 2 | 0

15. Secondary Outcome: Serum Neutralizing Anti-Toxin A and Anti-Toxin B Antibody Titers, as Measured by Toxin Neutralization Assay (TNA)
Description: Serum neutralizing anti-Toxin A and anti-Toxin B antibody titers are presented as Geometric Mean Titers (GMTs), as measured by TNA.
Time Frame: At Day 1, Day 31, Day 61, Day 180, Day 390, Day 491, Day 521 and Day 670
Population: The analysis was performed on the Per-Protocol Set for analysis of immunogenicity, which included all subjects who received one dose of the study treatment to which they were randomized and have post-vaccination immunogenicity data available at the specified time point, minus the subjects with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag 50 - 70 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | Placebo 50 - 70 Years Group
Number analyzed (Participants) | 9 | 10 | 45 | 42 | 29
Titer
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 1: number analyzed (Participants) | 9 | 10 | 35 | 31 | 19
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 1 | 7.24 [5.43 to 9.65] | 6.00 [6.00 to 6.00] | 6.00 [6.00 to 6.00] | 6.64 [5.70 to 7.72] | 6.25 [5.74 to 6.81]
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 31: number analyzed (Participants) | 9 | 10 | 35 | 31 | 19
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 31 | 55.52 [4.14 to 743.92] | 6.00 [6.00 to 6.00] | 8.87 [6.13 to 12.83] | 32.79 [16.34 to 65.80] | 6.74 [5.70 to 7.96]
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 61: number analyzed (Participants) | 8 | 10 | 35 | 31 | 19
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 61 | 108.68 [8.35 to 1414.69] | 6.00 [6.00 to 6.00] | 18.05 [10.54 to 30.93] | 407.04 [296.97 to 557.92] | 6.22 [5.76 to 6.72]
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 180 | 55.15 [6.32 to 481.00] | 6.00 [6.00 to 6.00] | 15.06 [10.17 to 22.32] | 207.62 [157.44 to 273.80] | 6.15 [5.85 to 6.45]
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 390: number analyzed (Participants) | 9 | 10 | 45 | 41 | 27
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 390 | 42.18 [5.16 to 344.79] | 6.00 [6.00 to 6.00] | 12.46 [8.86 to 17.52] | 101.46 [72.90 to 141.22] | 6.53 [5.73 to 7.45]
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 491: number analyzed (Participants) | 0 | 0 | 19 | 19 | 0
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 491 |  |  | 13.17 [7.76 to 22.36] | 73.63 [44.62 to 121.51] |
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 521: number analyzed (Participants) | 0 | 0 | 19 | 19 | 0
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 521 |  |  | 477.30 [204.95 to 1111.53] | 8276.96 [5290.84 to 12948.43] |
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 670: number analyzed (Participants) | 0 | 0 | 20 | 20 | 0
  Anti-toxin A neutralizing antibody titers/ HT-29, at Day 670 |  |  | 174.29 [92.64 to 327.90] | 1636.90 [1100.16 to 2435.51] |
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 1: number analyzed (Participants) | 9 | 10 | 35 | 31 | 19
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 1 | 9.26 [5.70 to 15.06] | 7.50 [7.50 to 7.50] | 9.17 [7.23 to 11.63] | 14.18 [8.79 to 22.88] | 8.31 [6.70 to 10.32]
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 31: number analyzed (Participants) | 9 | 10 | 35 | 31 | 19
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 31 | 50.11 [5.54 to 453.47] | 7.50 [7.50 to 7.50] | 23.61 [10.21 to 54.61] | 57.12 [19.16 to 170.24] | 8.83 [6.93 to 11.25]
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 61: number analyzed (Participants) | 9 | 10 | 35 | 27 | 19
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 61 | 42.68 [5.62 to 324.34] | 7.50 [7.50 to 7.50] | 27.67 [11.78 to 64.99] | 119.54 [41.49 to 344.42] | 8.73 [6.96 to 10.96]
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 180 | 35.92 [5.65 to 228.40] | 7.50 [7.50 to 7.50] | 21.08 [11.48 to 38.73] | 139.30 [74.75 to 259.60] | 9.35 [7.15 to 12.22]
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 390: number analyzed (Participants) | 9 | 10 | 45 | 41 | 27
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 390 | 28.93 [6.70 to 124.87] | 7.50 [7.50 to 7.50] | 18.24 [10.51 to 31.64] | 107.86 [60.93 to 190.93] | 9.30 [7.12 to 12.15]
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 491: number analyzed (Participants) | 0 | 0 | 19 | 19 | 0
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 491 |  |  | 37.00 [12.39 to 110.53] | 107.56 [39.93 to 289.77] |
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 521: number analyzed (Participants) | 0 | 0 | 19 | 17 | 0
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 521 |  |  | 207.45 [67.61 to 636.54] | 3590.97 [1468.26 to 8782.55] |
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 670: number analyzed (Participants) | 0 | 0 | 20 | 19 | 0
  Anti-toxin B neutralizing antibody titers/ HCT-116, at Day 670 |  |  | 101.18 [34.17 to 299.64] | 530.61 [212.57 to 1324.49] |
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 1: number analyzed (Participants) | 9 | 10 | 35 | 31 | 19
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 1 | 9.13 [5.80 to 14.37] | 7.50 [7.50 to 7.50] | 8.37 [7.12 to 9.83] | 11.71 [7.74 to 17.72] | 7.78 [7.20 to 8.40]
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 31: number analyzed (Participants) | 9 | 10 | 35 | 30 | 19
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 31 | 17.58 [5.97 to 51.76] | 7.50 [7.50 to 7.50] | 13.56 [8.37 to 21.99] | 20.86 [9.51 to 45.75] | 7.78 [7.20 to 8.40]
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 61: number analyzed (Participants) | 9 | 10 | 35 | 30 | 19
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 61 | 19.76 [5.28 to 74.00] | 7.50 [7.50 to 7.50] | 15.19 [8.89 to 25.96] | 20.61 [9.60 to 44.24] | 7.50 [7.50 to 7.50]
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 180 | 16.85 [6.59 to 43.04] | 7.50 [7.50 to 7.50] | 11.81 [8.29 to 16.81] | 20.63 [11.57 to 36.79] | 8.55 [6.98 to 10.49]
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 390: number analyzed (Participants) | 9 | 10 | 45 | 41 | 27
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 390 | 17.14 [5.70 to 51.56] | 7.50 [7.50 to 7.50] | 11.71 [8.26 to 16.60] | 19.00 [11.42 to 31.61] | 8.56 [6.95 to 10.55]
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 491: number analyzed (Participants) | 0 | 0 | 19 | 19 | 0
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 491 |  |  | 14.81 [7.31 to 30.01] | 17.21 [7.65 to 38.68] |
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 521: number analyzed (Participants) | 0 | 0 | 19 | 19 | 0
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 521 |  |  | 22.66 [8.92 to 57.61] | 34.48 [17.25 to 68.90] |
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 670: number analyzed (Participants) | 0 | 0 | 20 | 20 | 0
  Anti-toxin B neutralizing antibody titers/ IMR-90, at Day 670 |  |  | 19.57 [8.74 to 43.80] | 26.67 [13.10 to 54.30] |

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs were collected during the 7-day (Days 1-7) follow-up period after vaccination. Unsolicited AEs were collected during the 30-day (Day 1-30) follow-up period after vaccination. SAEs were collected from first vaccine dose (Day 1) up to study end (Day 670).
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe (within 30 days after any vaccine dose administration) according to occurrence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | CDIFF Ag 18 - 45 Years Group | Placebo 18 - 45 Years Group | CDIFF Ag + AS01B 50 - 70 Years Group | CDIFF Ag 50 - 70 Years Group | Placebo 50 - 70 Years Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/45 | 0/45 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 3/45 | 3/45 | 0/30
Other Adverse Events (participants affected / at risk) | 8/10 | 6/10 | 45/45 | 32/45 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDIFF Ag 18 - 45 Years Group (N=10) | Placebo 18 - 45 Years Group (N=10) | CDIFF Ag + AS01B 50 - 70 Years Group (N=45) | CDIFF Ag 50 - 70 Years Group (N=45) | Placebo 50 - 70 Years Group (N=30)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDIFF Ag 18 - 45 Years Group (N=10) | Placebo 18 - 45 Years Group (N=10) | CDIFF Ag + AS01B 50 - 70 Years Group (N=45) | CDIFF Ag 50 - 70 Years Group (N=45) | Placebo 50 - 70 Years Group (N=30)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 3 (3) | 15 (19) | 11 (11) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 21 (24) | 6 (6) | 6 (6)
Fatigue (General disorders) | 5 (5) | 2 (2) | 35 (47) | 14 (17) | 12 (14)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 20 (27) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 43 (78) | 2 (2) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 13 (15) | 6 (6) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 20 (26) | 6 (7) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dizziness exertional (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (4) | 25 (38) | 17 (23) | 9 (12)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT04026009/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04026009/SAP_001.pdf